CLINICAL TRIAL: NCT01854983
Title: Clinical Trial to Access Significance of Fluorescence Colposcopy With Autofluorescence Imaging for the Screening of Cervical Cancer
Brief Title: Significance of Fluorescence Colposcopy With Autofluorescence Imaging for Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jeong-Yeol Park, clinical assistant professor, Asan Medical Center
Other Study IDs: 2012-0693
Record Dates: First submitted 2013-05-14; First posted 2013-05-16 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Cervical Cancer
Keywords: fluorescence colposcopy; cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Clinical Trial to access Significance of fluorescence colposcopy with autofluorescence imaging for the screening of cervical cancer

DETAILED DESCRIPTION:
1. Perform pelvic vaginal exam of the subjective to know symptom, illness history, physical exam and basal state before fluorescence colposcopy.
2. Observe acetowhite epithelium and perform biopsy at suspicious lesion during fluorescence colposcopy.
3. Perform fluorescence colposcopy again after biopsy and confirm extraordinary reaction.
4. After 1~2weeks follow up the subjective at opd and confirm biopsy result.

ELIGIBILITY:
Inclusion Criteria:

1. age : 20-65 years
2. abnormal cervical papanicolaou smear , no other specific cervical disease
3. subject to colposcopic biopsy or LEEP
4. signed voluntarily to informed concents with full knowledge after explanation abot objective, method, contents

Exclusion Criteria:

1. pregnant women
2. porphyria
3. severe cervical bleeding
4. genital chlamydia, gonorrhea infection
5. other drug user with possible interaction (e.g. photosensitizer)
6. no informed consent

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: tertiary center
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
fluorescence colposcopic result | 2weeks after fluorescence colposcopy

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Yeol Park, M.D., Ph.D., Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea